CLINICAL TRIAL: NCT00935480
Title: IMPACT OF THERAPY INTENSIFICATION BY AN INTEGRASE INHIBITOR +/- CCR5 INHIBITOR ON THE LYMPHOID RESERVOIR FOR HIV-1 IN CHRONICALLY INFECTED PATIENTS
Brief Title: IntensVIH: Impact Of Therapy Intensification By An Integrase Inhibitor +/- CCR5 Inhibitor On The Lymphoid Reservoir For Hiv-1 In Chronically Infected Patients
Acronym: IntensVIH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-2009.01
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: HIV Infections
Keywords: HIV; INTEGRASE INHIBITOR; Inhibitor on the lymphoid reservoir; Residual HIV replication; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAART+Raltegravir 12 months (+/-) Maraviroc (Experimental)
  Interventions: Drug: Isentress®; Drug: Celsentri®
- HAART (No Intervention)

INTERVENTIONS:
Drug: Isentress® — P.O, 1 tablet containing 400 mg every 12 hours
  Arms: HAART+Raltegravir 12 months (+/-) Maraviroc
Drug: Celsentri® — p.o.: 1 tablet containing 150 mg morning and evening (due to combination with PI/r) or containing 300 mg if fosamprenavir/r is used as the PI (MA)
  Arms: HAART+Raltegravir 12 months (+/-) Maraviroc

SUMMARY:
To determine the efficacy of adding Isentress®, with or without Celsentri®, to effective conventional antiretroviral therapy (comprising at least 2 reverse transcriptase inhibitors and one boosted protease inhibitor), on residual HIV replication and blood cell and gut-associated lymphoid tissue reservoirs (reverse transcriptase inhibitors: RTIs, boosted protease inhibitors: PI/r).

To evaluate the effect of therapy intensification by means of an integrase inhibitor with or without CCR5 inhibitor treatment on the lymphoid reservoir in patients chronically infected with HIV-1, successfully treated with "conventional triple therapy", measured by:

* residual plasma replication between 0 and 50 copies/ml
* intracellular HIV RNA levels in circulating lymphocytes (PBMC) and lymphocytes in gut-associated rectal lymphoid tissue (RL).
* proviral HIV DNA levels in PBMC and RL.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged over 18 years
* HIV infection confirmed by Western Blot
* Karnofsky score > 80%
* Treatment-experienced patients having received combined antiretroviral therapy including at least 2 RTI and 1 PI/r for at least 12 months with plasma viral load <50 copies/ml for at least 6 months
* Stable first-line treatment (or other, if changes were not made for reasons relating to viral resistance) with 2 RTIs and 1 PI/r
* Proper safety and compliance for the ongoing combination;
* Patient agreeing to undergo 3 proctosigmoidoscopy examinations over a 12-month period;
* Plasma HIV-1 RNA <50 copies/ml at inclusion;
* Circulating CD4 >200/mm3 at inclusion;
* Isentress® and Celsentri®-naïve patients
* No contraindications to the use of the investigational products
* Written, informed consent, obtained from the patient or his/her legal representative.

Exclusion Criteria:

1. Opportunistic infection or active tumor disease
2. Chronic diarrhea, malabsorption, progressive enteric infection
3. Aged under 18 years
4. Pregnancy - breast-feeding ( a pregnancy test will be done at the inclusion visit)
5. Co-infection with HIV-2
6. History of immunomodulator treatment (interleukin-2, alpha-interferon)
7. Ongoing treatment of HBV or HCV co-infection
8. Blood constitution disorders
9. Contraindications to the administration of raltegravir or maraviroc
10. Circulating CD4 nadir <100/mm3 in the natural history of HIV-1 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2010-11-12 (Actual); Study Completion 2014-08-08 (Actual)

PRIMARY OUTCOMES:
residual plasma replication between 0 and 50 copies/ml | one year
intracellular HIV RNA levels in circulating lymphocytes (PBMC) and lymphocytes in gut-associated rectal lymphoid tissue (RL | one year
proviral HIV DNA levels in PBMC and RL | one year

SECONDARY OUTCOMES:
CD4 counts | one year
CD8 activation levels | one year

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer, Service d'infectiologie, Toulon
  - Centre Hospitalier Intercommunal de Toulon La Seyne sur mer, Toulon

REFERENCES:
- [Derived] Lafeuillade A, Assi A, Poggi C, Bresson-Cuquemelle C, Jullian E, Tamalet C. Failure of combined antiretroviral therapy intensification with maraviroc and raltegravir in chronically HIV-1 infected patients to reduce the viral reservoir: the IntensHIV randomized trial. AIDS Res Ther. 2014 Oct 7;11(1):33. doi: 10.1186/1742-6405-11-33. eCollection 2014. PMID 25320633